CLINICAL TRIAL: NCT03342118
Title: Effect of Oral Phloroglucin (Flospan®) as Premedication of Non-sedative Diagnostic Esophagogastroduodenoscopy: Single Center, Prospective, Double Blinded, Randomized Controlled Trial
Brief Title: Effect of Oral Phloroglucin (Flospan®) as Premedication of Non-sedative Diagnostic Esophagogastroduodenoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, YooJin Lee, Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-06-043
Record Dates: First submitted 2017-08-16; First posted 2017-11-14 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Anti-spasmodics; Gastric Peristalsis; Non-sedative Endoscopy
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phloroglucin group (Experimental): patients taken Phloroglucin(Flospan®)
  Interventions: Drug: Phloroglucin(Flospan®)
- Normal saline placebo group (Placebo Comparator): patients taken normal saline placebo
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Phloroglucin(Flospan®) — The experimental group was taken with Phloroglucin(Flospan®) before endoscopy.
  Arms: Phloroglucin group
Drug: Normal saline — The control group was treated with normal saline before endoscopy
  Arms: Normal saline placebo group

SUMMARY:
Gastric peristalsis, which occurs during the endoscopic procedure, limits the visual inspection of the inspection field, causing interference in the inspection. The actual endoscopic examination is most commonly used by injecting Hyoscine butylbromide(Buscopan®), Cimetropium bromide (Algiron ®) into intravenous or muscular injection so it is not suitable for patients who undergo non-sedative esophagogastroduodenoscopy. In addition, these drugs were reported the side effects including thirst, dysuria, transient visual filed defect, tachycardia, anxiety so were not recommended for benign prostate hyperplasia, glaucoma, old age patients. For comfort and succesfull test, anti-spasmodics which don't have anti-cholinergic effect and are possible to take orally is necessary. Phloroglucin(Flospan®) is a smooth muscle relaxant that is currently used in the anti-spasmodic treatment without anticholinergic action so it can be administered in patients with glaucoma or BPH. Also it is suitable for endoscopic premedication due to transparent liquid component. Therefore, in this study, we would like to confirm the efficacy and safety of Phloroglucin (Flospan ®), which can be taken orally, as an pre-medication for non-sedative endoscopy.

DETAILED DESCRIPTION:
Background : Endoscopy is currently widely regarded as the most important test in diagnosing stomach disorders, including stomach cancer. Gastric peristalsis, which occurs during the endoscopic procedure, limits the visual filed of the inspection, causing interference in the inspection. The actual endoscopic examination is most commonly used by injecting Hyoscine butylbromide(Buscopan®), Cimetropium bromide (Algiron ®) into intravenous or muscular injection so it is not suitable for patients who undergo non-sedative endoscopy because intravenous assessment is unnecessary. In addition, these drugs were reported the side effects including thirst, dysuria, transient visual filed defect, tachycardia, anxiety so were not recommended for patients with benign prostatic hyperplasia, glaucoma, old age. Actually patients who undergo non-sedative endoscopy are used to perform examinations without using anti-spasmodics. In this case, gastric peristalsis restricts endoscopist's visibility and making accurate observation and prolonged inspection time increases patient's discomfort. For comfort and successfull test, anti-spasmodics which don't have anti-cholinergic effect and are possible to take orally is necessary. Phloroglucin(Flospan®) prompts to release norepinephrine by impeding catecholamine O-methyl transferase enzymes in visceral smooth muscle, so it works to control spasm by normalizing smooth muscle movement which was accelerated by acetylcholine. Phloroglucin(Flospan®) is a smooth muscle relaxant that is currently used in the anti-spasmodic treatment without anticholinergic action so it can be administered in patients with glaucoma or BPH. Also it is suitable for endoscopic premedication due to transparent liquid component. Therefore, in this study, we would like to confirm the efficacy and safety of Phloroglucin (Flospan ®), which can be taken orally, as an pre-medication for non-sedative endoscopy.

Aim : Analysis for the effects of Phloroglucin (Flospan ®) as pre-medication for non-sedative endoscopy

Material and methods : This study is a single center, prospective, double blinded, randomized controlled trial that will be performed in Keimyung University Dongsan medical center. A total of 134 patients aged 18 to 80 are enrolled and patients were randomly assigned to the test group and the placebo group, taking the test drug or placebo 10 minutes before the endoscopy. The endoscopist records the degree of peristaltic movement and the degree of difficulty of the test at the start and end of the test. The degree of the peristalsis and the discomfort of the examination are evaluated by the scale used in the previous study. The questionnaire will be used to evaluate the patient's discomfort after drug administration, the taste of the drug, and the intention to re-use the drug.

ELIGIBILITY:
Inclusion Criteria:

* patients who perform non-sedative endoscopy for diagnosis or screening purposes.
* patients who understand and follow the directions and questionnaires of clinical trials.
* patients who have decided to voluntarily participate in this clinical trial and have agreed in writing

Exclusion Criteria:

* Patients who performed Upper GI surgery.
* Severe gastric outlet obstruction or malformations or gastroparesis
* Patients who have severe cognitive impairment
* Pregnant or lactation patients
* Patients who need to hemostasis for upper GI bleeding
* Hemodynamic unstable patients
* Above American Society of Anesthesiology classification class 4

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
Peristasis changes from baseline at the moment of endoscopy | 1day
  Modified peristalsis grade (No, weak, moderate, severe, very severe)

SECONDARY OUTCOMES:
Discomfort of endoscopy | 1day
  Simplified discomfort grade questionnaire (Very easy, easy, so so, difficult)
Taste of the drug | 1day
  Taste grade (Poor, bad, so so, good, very good)

CONTACTS AND LOCATIONS:
Locations (1):
- KeimyungUniversity, Daegu, Jung-gu, South Korea

REFERENCES:
- [Derived] Jung H, Kim HJ, Choi ES, Lee JY, Park KS, Cho KB, Lee YJ. Effectiveness of oral phloroglucinol as a premedication for unsedated esophagogastroduodenoscopy: A prospective, double-blinded, placebo-controlled, randomized trial. PLoS One. 2021 Aug 4;16(8):e0255016. doi: 10.1371/journal.pone.0255016. eCollection 2021. PMID 34347808